CLINICAL TRIAL: NCT00478244
Title: Allogeneic Hematopoietic Cell Transplantation to Correct the Biochemical Defect and Create Tolerance to Donor Tissue in Subjects With Epidermolysis Bullosa
Brief Title: Allogeneic Hematopoietic Stem Cell Transplant For Epidermolysis Bullosa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Competing studies
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2006-15; CDR0000546620 (Other: PDQ); UMN-0702M01504 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Epidermolysis Bullosa
Keywords: epidermolysis bullosa; dystrophic epidermolysis bullosa
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica | interventions — Busulfan; Cyclophosphamide; fludarabine phosphate; fludarabine; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epidermolysis Bullosa (EB) Patients (Experimental): Epidermolysis bullosa patients treated per study regimen with chemotherapy and stem cell transplant.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Procedure: hematopoietic bone marrow transplantation

INTERVENTIONS:
Drug: busulfan — Day -9 through Day -6: 1.1 mg/kg if < 12 kg IV every 6 hours; 0.8 mg/kg if > 12 kg.
  Other Names: Bulsulfex
Drug: cyclophosphamide — Day -5 through Day -2: 50 mg/kg IV over 120 min.
  Other Names: Cytoxan
Drug: fludarabine phosphate — Day -5 through Day -3: 25 mg/m2 IV over 60 min.
  Other Names: Fludarabine; Fludara
Procedure: hematopoietic bone marrow transplantation — allogeneic bone marrow, peripheral stem cell or umbilical cord blood transplantation
  Other Names: Bone marrow transplant

SUMMARY:
RATIONALE: In animal models, stem cells have been shown to home to the skin and repair the biochemical and structural abnormalities associated with recessive dystrophic epidermolysis bullosa (RDEB) (collagen 7 deficiency).

PURPOSE: To determine the safety and effectiveness of stem cell infusion in the treatment of RDEB.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the incidence of detectable donor-derived collagen type VII at day 100 in patients with epidermolysis bullosa by donor.

Secondary

* Determine the incidence of transplant-related mortality at day 180
* Determine the incidence of blood chimerism at days 21, 100, 180, 365, and 730
* Determine the incidence of neutrophil recovery at day 42 and platelet recovery at day 180
* Determine the incidence of acute graft-versus-host disease (GVHD) grade II-IV and grade III-IV at day 100
* Determine the incidence of chronic GVHD at 1 year
* Determine the probability of survival at 1 and 2 years
* Determine the incidence of donor derived cells in the skin
* Determine resistance to blister formation OUTLINE: This is an open-label, pilot study.
* Conditioning regimen: Busulfan intravenously (IV) over 2 hours every 6 hours on days -9 to -4, fludarabine phosphate IV over 1 hour on days -5 to -3, and high-dose cyclophosphamide IV over 1 hour on days -5 to -2.
* Stem cell transplantation on day 0.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: 30 patients

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of epidermolysis bullosa (EB)

  * Documented collagen type VII deficiency by:

    * Antigenic mapping (LH7.2 antibody)
    * Ultrastructure analysis of anchoring fibrils
    * DNA mutation analysis
* Performance status: >50% Lansky; >50% Karnofsky
* Adequate organ function

  * Renal: glomerular filtration rate > 60ml/min/1.73m2 patients aged ≤ 10 years
  * Hepatic: bilirubin, aspartate aminotransferase/alanine aminotransferase (AST/ALT), Alkaline phosphatase (ALP) < 5 x upper limit of normal 4.2.3 Pulmonary: oxygen saturation >92% 4.2.4 Cardiac: left ventricular ejection fraction > 45%.
* Healthy related hematopoietic stem cell donor available and meeting 1 of the following criteria:

  * HLA-A, B, DRB1-identical sibling bone marrow and/or umbilical cord blood donor (first priority)
  * HLA-A, B, DRB1-matched or partially matched related donor (second priority)
  * Donor may be a carrier but must be unaffected by EB
  * 8/8 HLA A, B, C, DRB1 allele level matched unrelated marrow donor (third priority)
  * 7/8 HLA-A, B, C, DRB1 allele level matched unrelated marrow donor or 4/6 HLA-A, B (antigen level), DRB1 (allele level) matched unrelated cord blood donor (fourth priority)

Exclusion criteria:

* Active infection at time of transplantation (including active infection with Aspergillus or other mold within 30 days)
* Squamous cell carcinoma of the skin
* History of human immunodeficiency virus (HIV) infection
* Prior transplantation with donor skin

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2007-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Wagner, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Wagner JE, Ishida-Yamamoto A, McGrath JA, Hordinsky M, Keene DR, Woodley DT, Chen M, Riddle MJ, Osborn MJ, Lund T, Dolan M, Blazar BR, Tolar J. Bone marrow transplantation for recessive dystrophic epidermolysis bullosa. N Engl J Med. 2010 Aug 12;363(7):629-39. doi: 10.1056/NEJMoa0910501. PMID 20818854

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were registered with the BMT Biostatistical Support Group at the University of Minnesota.
Groups:
- Epidermolysis Bullosa (EB) Patients: Epidermolysis bullosa patients enrolled for treatment with chemotherapy (Busulfan 0.8 or 1.1 mg/kg Days 6-9 before transplant; Fludarabine 25 mg/m^2 Days 3-5 before transplant; Cyclophosphamide 50 mg/kg Days 2-5 before transplant) and stem cell infusion (Day 0) followed by donor epidermal transplant .
Period: Overall Study
Arm/Group | Epidermolysis Bullosa (EB) Patients
Started | 7
Completed | 6
Not Completed | 1
Not completed — Did not receive transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Epidermolysis Bullosa (EB) Patients
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With >70% Donor Chimerism
Description: Number of patients with donor chimerism - percentage of donor cells in the patient via the peripheral blood or bone marrow.
Time Frame: Days 21, 100, 180, 365 and 730 Post Transplant
Measure: Number; unit: participants
Groups:
- Evaluable Patients: Includes only patients that received transplant (one patient died prior to transplant).
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants
  Day 21 | 6
  Day 100 | 5
  Day 180 | 5
  Day 365 | 5
  Day 730 | 5

2. Secondary Outcome: Number of Patients With Transplant-Related Mortality
Description: Number of patients who died due to complications of the transplant (includes all deaths without previous relapse or progression).
Time Frame: Day 180 Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants | 0

3. Secondary Outcome: Number of Patients With Platelet Engraftment
Description: Number of patients with a platelet count >5 x 10^10 cells/liter for 3 consecutive measurements.
Time Frame: Day 180 Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants | 5

4. Secondary Outcome: Number of Patients With Acute Graft-Versus-Host Disease (GVHD)
Description: Number of patients with GVHD. Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Time Frame: Day 100 Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants | 1

5. Secondary Outcome: Number of Patients With Chronic Graft-Versus-Host Disease (cGVHD)
Description: Number of patients with cGVHD; a severe long-term complication created by infusion of donor cells into a foreign host.
Time Frame: Day 365 Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants | 0

6. Secondary Outcome: Overall Survival
Description: Survival is defined as the number of patients that were alive post transplant.
Time Frame: 1 year and 2 years Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants
  1 Year Post Transplant | 5
  2 Years Post Transplant | 5

7. Secondary Outcome: Number of Patients With Donor Derived Cells in Skin
Description: Number of patients who had donor skin chimerism - donor cells in the patient's epidermis (a state in bone marrow transplantation in which bone marrow and host cells exist compatibly without signs of graft-versus-host rejection disease).
Time Frame: Day 90 Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants | 6

8. Secondary Outcome: Number of Patients With Resistance to Blister Formation
Description: Resistance to Blister Formation demonstrated by response to negative pressure.
Time Frame: Month 1 through Month 24 Inclusive
Population: Added blister formation testing later in study; only 2 patients had pre-transplant test.
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 2
participants | 2

9. Secondary Outcome: Number of Patients With Neutrophil Engraftment
Description: Number of patients with an absolute neutrophil count >5 x 10^8 cells/liter for 3 consecutive days.
Time Frame: Day 42 Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants | 6

10. Primary Outcome: Number of Patients With Detectable Collagen Type VII
Description: Number of patients with epidermolysis bullosa who had collagen type VII. Type VII collagen defects cause recessive dystrophic epidermolysis bullosa (RDEB), a blistering skin disorder often accompanied by epidermal cancers.
Time Frame: Day 100 Post Transplant
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 6
participants | 5

ADVERSE EVENTS:
Time Frame: All subjects were monitored continuously and only serious unexpected and selected serious adverse experiences were collected during the first 100 days after cell infusion.
Description: Serious adverse events include: marrow engraftment failure, severe acute graft-versus-host (GVHD) (Grades III and IV), and death. Death was collected on 6 of 7 patients enrolled.
Arm/Group | Epidermolysis Bullosa (EB) Patients
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidermolysis Bullosa (EB) Patients (N=7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 6 (6)
Death (General disorders) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2) — Candida sepsis
Grade IV skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1)
Graft failure (Blood and lymphatic system disorders) | 1 (1)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 4 (4)
Renal insufficiency (Renal and urinary disorders) | 2 (2)
Viral infection (Infections and infestations) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes